CLINICAL TRIAL: NCT01983046
Title: The Effects of Rectal Administration of SCFA on Human Substrate and Energy Metabolism
Brief Title: Rectal Short Chain Fatty Acids Combinations and Substrate and Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: NL44507.068
Record Dates: First submitted 2013-09-17; First posted 2013-11-13 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Obesity; Type 2 Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Butyrates; Propionates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Three different mixture of acetate, butyrate and propionate and palcebo
- high acetate ratio (Active Comparator): high acetate ratio
  Interventions: Drug: Three different mixture of acetate, butyrate and propionate and palcebo
- high butyrate ratio (Active Comparator): high butyrate ratio
  Interventions: Drug: Three different mixture of acetate, butyrate and propionate and palcebo
- high propionate ratio (Active Comparator): high propionate ratio
  Interventions: Drug: Three different mixture of acetate, butyrate and propionate and palcebo

INTERVENTIONS:
Drug: Three different mixture of acetate, butyrate and propionate and palcebo

SUMMARY:
Gut microbiota is being increasingly recognized as an important factor in fat distribution, insulin sensitivity and glucose and lipid metabolism. Accordingly, the intestinal microbiota could play an important role in the development of obesity and type 2 diabetes mellitus. The role of gut-derived short-chain fatty acids (SCFA), the formation of which is enhanced by microbial fermentation of fiber, is still controversial. One study found that an increase in the formation of SCFA stimulated energy extraction from diet, with subsequent weight gain. In contrast, supplementation of non-fermentable carbohydrates, which lead to an increase in SCFA formation, had beneficial effects on body weight control and insulin sensitivity. Of note, a study showed that butyrate supplementation in mice prevented diet-induced obesity and insulin resistance. At the present time, our understanding of the effects of SCFA on human metabolism (in gut or systemically) is still limited. Yet, in light of the health claims of certain dietary fibers (prebiotics), a detailed picture of the physiology of human SCFA metabolism and its interaction with the microbiome is of pivotal importance. We hypothesize that the differential availability of SCFA impacts human metabolism differently. To determine whether rectal administration of SCFA is a good model for studying the metabolic effects of SCFA we first have performed a pilot study (METC 11-3-079). In this pilot study we have determined if rectal administration of sodium acetate has the same effects on substrate and energy metabolism compared to proximal administration. Our results indicate that the primary outcome parameter fat oxidation was significantly changed during post-absorptive conditions, when sodium acetate in a concentration of 180mM was administered in the distal part of the colon. In contrast, no effect on energy expenditure or substrate oxidation was seen when sodium acetate was administered in the proximal colon. Consequently, the distal part of the colon seems to be a good model to determine effects of gut-derived SCFA on the human substrate and energy metabolism. Therefore, we will administer in this study the SCFA rectally by using enemas. We will administer different combinations of SCFA to healthy, overweight male volunteers and examine effects on metabolism. This study is an important part of a Gastrointestinal Health TIFN project (GH003 WP 1.2), which will provide more insight in how increased availability of a beneficial SCFA mixture might serve as a basis for rational nutritional strategies in the prevention and treatment of obesity and type 2 diabetes mellitus. To obtain rational nutritional strategies, a next step in this TIFN project will be focusing on dietary ingredients modulating intestinal microbiota and subsequent SCFA production.

ELIGIBILITY:
Inclusion Criteria:

* Overweight
* Obese men

Exclusion Criteria:

* Athletes
* Diabetes mellitus

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
fat oxidation | 4 hours total (2 hours fasting, 2 hours postprandial)
  we will measure fat oxidation and energy expenditure by using the ventilated hood system

SECONDARY OUTCOMES:
Hormones that influence energy metabolism | 4 hours total (2 hours fasting and 2 hours postprandial)
Circulating metabolites | 4 hours total (2 hours fasting and 2 hours postprandial)
Hormones that influence energy metabolism - Circulating metabolites - Inflammatory markers - plasma SCFA content; - Indirect markers of insulin sensitivity - Appetite (VAS-scoring). | 4 hours total (2 hours fasting and 2 hours postprandial)

CONTACTS AND LOCATIONS:
Locations (1):
- University Maastricht, Maastricht, Limburg, Netherlands